CLINICAL TRIAL: NCT04503551
Title: A Phase III, Multicenter, Randomized Study of the Efficacy, Safety, and Pharmacokinetics of the Port Delivery System With Ranibizumab in Patients With Diabetic Retinopathy
Brief Title: A Multicenter, Randomized Study in Participants With Diabetic Retinopathy Without Center-involved Diabetic Macular Edema To Evaluate the Efficacy, Safety, and Pharmacokinetics of Ranibizumab Delivered Via the Port Delivery System Relative to the Comparator Arm
Acronym: PAVILION
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GR41675
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Results first posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Retinopathy
Keywords: Port Delivery System; ranibizumab; Diabetic Retinopathy; anti-VEGF, nonproliferative diabetic retinopathy, retina, vision loss, retinal disease, eye disease
MeSH Terms: conditions — Diabetic Retinopathy; Vision Disorders; Retinal Diseases; Eye Diseases | interventions — Ranibizumab; Injections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The visual acuity examiner will only conduct refraction and visual acuity assessments and will be masked, as best as possible, to the following items: study eye assignment; study visit type; and treatment assignment.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PDS Arm (Experimental): Participants randomized to the PDS arm will receive two intravitreal ranibizumab injections and will then have the PDS implant (pre-filled with ranibizumab) surgically inserted. PDS implant refill-exchange procedures will be performed on a fixed interval every 36-weeks (Q36W) thereafter
  Interventions: Drug: PDS Implant Pre-Filled with 100 mg/mL Ranibizumab; Drug: Intravitreal Ranibizumab 0.5 mg Injection
- Comparator Arm (Other): Participants randomized to the comparator arm will undergo study visits every 4 weeks (Q4W) for comprehensive clinical monitoring until they receive the PDS implant (pre-filled with ranibizumab). PDS implant refill-exchange procedures will be performed on a fixed interval Q36W thereafter. Participants will be eligible to receive intravitreal ranibizumab 0.5 mg injections if treatment eligibility criteria are met.
  Interventions: Drug: PDS Implant Pre-Filled with 100 mg/mL Ranibizumab; Drug: Intravitreal Ranibizumab 0.5 mg Injection

INTERVENTIONS:
Drug: PDS Implant Pre-Filled with 100 mg/mL Ranibizumab — Will be administered as per the schedule described in individual arm.
Drug: Intravitreal Ranibizumab 0.5 mg Injection — Will be administered as per the schedule described in individual arm.

SUMMARY:
Study GR41675 is a Multicenter, Randomized Study in Participants with Diabetic Retinopathy (DR) Without Center-Involved Diabetic Macular Edema (CI-DME) to Evaluate the Efficacy, Safety of the Port Delivery System with Ranibizumab (PDS) Relative to the Comparator Arm

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at time of signing Informed Consent Form
* Documented diagnosis of diabetes mellitus (Type 1 or Type 2)
* HbA1c level of ≤12% within 2 months prior to screening or at screening

Inclusion Criteria for Study Eye

* Moderately severe or severe NPDR (ETDRS-DRSS level 47 or 53)
* BCVA score of ≥ 69 letters (20/40 approximate Snellen equivalent or better)

Exclusion Criteria:

* Uncontrolled blood pressure
* Cerebrovascular accident or myocardial infarction within 6 months prior to randomization
* Atrial fibrillation diagnosis or worsening within 6 months prior to randomization
* Current systemic treatment for a confirmed active systemic infection
* Renal failure requiring renal transplant, hemodialysis, or peritoneal dialysis, or anticipated to require hemodialysis or peritoneal dialysis at any time during the study
* History of other disease, other non-diabetic metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a condition that contraindicates the use of ranibizumab or surgical placement of the PDS implant; that might affect interpretation of the results of the study; or that renders the patient at high risk for treatment complications in the opinion of the investigator or Sponsor

Ocular Exclusion Criteria for Study Eye:

* Presence of center-involved diabetic macular edema (defined as CST ≥325 µm)
* Any intravitreal anti-VEGF treatment at any time prior to randomization
* Any use of medicated intraocular implants, including Ozurdex® or Iluvien® implants at any time prior to randomization
* Any intravitreal corticosteroid treatment at any time prior to randomization
* Any periocular (e.g., subtenon) corticosteroid treatment at any time prior to randomization
* Any PRP at any time prior to randomization
* Any macular laser photocoagulation (such as micropulse and focal or grid laser) at any time prior to randomization
* Active intraocular inflammation (grade trace or above)
* Clinically significant abnormalities of the vitreous-retinal interface involving the macular area or disrupting the macular architecture, such as vitreous-retinal traction or epiretinal membrane (assessed by the investigator and confirmed by the central reading center)
* Uncontrolled ocular hypertension or glaucoma and any such condition the investigator determines may require a glaucoma-filtering surgery during a participant's participation in the study
* History of glaucoma-filtering surgery, tube shunts, or microinvasive glaucoma surgery
* Any concurrent ocular condition (e.g., cataract, epiretinal membrane) that would require surgical intervention during the study to prevent or treat visual loss that might result from that condition
* Any concurrent ocular condition (e.g., amblyopia, strabismus) that may affect interpretation of study results
* History of other ocular diseases that gives reasonable suspicion of a disease or condition that contraindicates the use of ranibizumab, that might affect interpretation of study results, or that renders the participant at high risk for treatment complications

Ocular Exclusion Criteria for Either Eye

* Suspected or active ocular or periocular infection of either eye
* Any history uveitis including idiopathic, drug-associated or autoimmune-associated uveitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2026-01-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (64):
- United States (63):
  - Barnet Dulaney Perkins Eye Center, Mesa, Arizona
  - Retinal Consultants of Arizona;Opthalmology, Phoenix, Arizona
  - Associated Retina Consultants, Phoenix, Arizona
  - California Retina Consultants, Bakersfield, California
  - The Retina Partners, Encino, California
  - Retina Consultants of Orange County;Clinical Research, Fullerton, California
  - Jules Stein Eye Institute/ UCLA, Los Angeles, California
  - California Eye Specialists Medical Group, Pasadena, California
  - Kaiser Permanente;RESEARCH AND EVALUATION, Riverside, California
  - Retina Consultants Medical Group, Sacramento, California
  - Orange County Retina Medical Group, Santa Ana, California
  - Southwest Retina Research Center, Durango, Colorado
  - Colorado Clinical Research, Lakewood, Colorado
  - Retina Group of New England, Waterford, Connecticut
  - Retina Specialty Institute, Pensacola, Florida
  - Fort Lauderdale Eye Institute, Plantation, Florida
  - Retina Associates of Florida;Retina Associates of Florida, Tampa, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Georgia Retina, Marietta, Georgia
  - Retina Consultants of Hawaii at Pali Momi Medical Center, ‘Aiea, Hawaii
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Illinois Retina Associates, Joliet, Illinois
  - University Retina, Lemont, Illinois
  - Retina Associates, Lenexa, Kansas
  - Maine Eye Center, Portland, Maine
  - The Retina Care Center, Baltimore, Maryland
  - Johns Hopkins Hospital;Johns Hopkins Med;Wilmer Eye Inst, Baltimore, Maryland
  - Cumberland Valley Retina Consultants;Clinical Research, Hagerstown, Maryland
  - Associated Retinal Consultants - Royal Oak, Royal Oak, Michigan
  - VitreoRetinal Surgery PLLC;DBA Retina Consultants of Minnesota, Minneapolis, Minnesota
  - Pepose Vision Institute, Chesterfield, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - Envision Ocular, LLC, Bloomfield, New Jersey
  - Retina Associates of New Jersey, Teaneck, New Jersey
  - Retina Vitreous Surgeons of Central New York, Liverpool, New York
  - New York University (NYU), New York, New York
  - Asheville Eye Associates Western Carolina Retinal Associates;Clinical Research, Asheville, North Carolina
  - Charlotte Eye Ear Nose and Throat Associates- SouthPark;Retina, Charlotte, North Carolina
  - Duke Eye Center, Durham, North Carolina
  - Cape Fear Retinal Associates, Wilmington, North Carolina
  - Ohio State Havener Eye Institute;Ophthalmology Research, Columbus, Ohio
  - Retina Vitreous Center - Glen Eagles, Edmond, Oklahoma
  - Retina Northwest;Research Department, Portland, Oregon
  - Mid Atlantic Retina;Retina Research, Philadelphia, Pennsylvania
  - Charleston Neuroscience, Ladson, South Carolina
  - Palmetto Retina Center, West Columbia, South Carolina
  - Charles Retina Institution;Retina surgery, Germantown, Tennessee
  - Southeastern Retina Associates, Knoxville, Tennessee
  - Tennessee Retina, Nashville, Tennessee
  - Retina Research Institute of Texas, Abilene, Texas
  - Austin Retina Associates;Opthalmology, Austin, Texas
  - Retina & Vitreous of Texas, Bellaire, Texas
  - Texas Retina Associates;Research, Dallas, Texas
  - Retina Center of Texas, Grapevine, Texas
  - Retina Consultants of Texas, Houston, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Rocky Mountain Retina Consultants, Murray, Utah
  - Retina Associates of Utah, PLLC;Clinical Research, Salt Lake City, Utah
  - Piedmont Eye Center, Lynchburg, Virginia
  - Wagner Kapoor Institute;Opthalmology, Norfolk, Virginia
  - Retina Institute of Virginia, Richmond, Virginia
  - Pacific Northwest Retina, Silverdale, Washington
  - Spokane Eye Clinical Research;Spokane Eye Surgery Center, Spokane, Washington
- Emanuelli Research & Development Center, Arecibo, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Pieramici DJ, Awh CC, Chang M, Emanuelli A, Holekamp NM, Hu AY, Suner IJ, Wykoff CC, Brittain C, Howard D, Quezada-Ruiz C, Santhanakrishnan A, Latkany P. Port Delivery System With Ranibizumab vs Monitoring in Nonproliferative Diabetic Retinopathy Without Macular Edema: The Pavilion Randomized Clinical Trial. JAMA Ophthalmol. 2025 Apr 1;143(4):317-325. doi: 10.1001/jamaophthalmol.2025.0001. PMID 40048178

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in this study at 50 investigative sites in the United States from 10 August 2020. The study is ongoing. The analyses presented in this results summary are based on a primary completion date (clinical cut-off) of 03 October 2022.
Pre-assignment Details: A total of 174 participants with moderately severe or severe non-proliferative diabetic retinopathy (NPDR) without center-involved diabetic macular edema (CI-DME) were randomized in a 5:3 ratio to either port delivery system (PDS) arm or comparator arm.
Groups:
- PDS With Ranibizumab 100 mg/mL: Participants received two loading doses of ranibizumab, 0.5 mg, as IVT before the PDS implant procedure. The first loading dose was on Day 1 followed by the second dose at Week 4. The PDS implant (pre-filled with ranibizumab 100 mg/mL) was surgically inserted 1 to 14 days after the second loading dose. Participants underwent PDS implant refill-exchange procedures (ranibizumab 100 mg/mL) Q36W thereafter until the end of study.
- Comparator Arm: Participants underwent study visits every 4 weeks (Q4W) for observation and comprehensive clinical monitoring for the first 60 weeks. Thereafter, participants received two loading doses of ranibizumab, 0.5 mg, as IVT before the PDS implant procedure. The first loading dose was scheduled at Week 60 followed by the second dose at Week 64. The PDS implant (pre-filled with ranibizumab 100 mg/mL) was surgically inserted 1 to 14 days after the second loading dose. Participants underwent PDS implant refill-exchange procedures (ranibizumab 100 mg/mL) Q36W thereafter until the end of study.
Period: Overall Study
Arm/Group | PDS With Ranibizumab 100 mg/mL | Comparator Arm
Started | 106 | 68
Safety Evaluable Population (Safety Evaluable Population included all participants who received any study treatment, and participants randomized to the comparator arm under observation, grouped according to treatment actually received prior to Week 52.) | 105 | 68
Completed | 0 | 0
Not Completed | 106 | 68
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Physician Decision | 1 | 0
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — Ongoing at Week 52 | 99 | 62

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) Population included all participants who were randomized. Participants were grouped according to treatment assigned at randomization.
Groups:
- Comparator Arm: Participants underwent study visits Q4W for observation and comprehensive clinical monitoring for the first 60 weeks. Thereafter, participants received two loading doses of ranibizumab, 0.5 mg, as IVT before the PDS implant procedure. The first loading dose was scheduled at Week 60 followed by the second dose at Week 64. The PDS implant (pre-filled with ranibizumab 100 mg/mL) was surgically inserted 1 to 14 days after the second loading dose. Participants underwent PDS implant refill-exchange procedures (ranibizumab 100 mg/mL) Q36W thereafter until the end of study.
- Total: Total of all reporting groups
Arm/Group | PDS With Ranibizumab 100 mg/mL | Comparator Arm | Total
Number analyzed (Participants) | 106 | 68 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (11.32) | 54.1 (12.30) | 53.9 (11.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 27 | 74
  Male | 59 | 41 | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 29 | 72
  Not Hispanic or Latino | 63 | 39 | 102
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 0 | 4
  Asian | 9 | 8 | 17
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 14 | 4 | 18
  White | 73 | 52 | 125
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a ≥2-Step Improvement From Baseline on the Early Treatment Diabetic Retinopathy Study-Diabetic Retinopathy Severity Scale (ETDRS-DRSS) at Week 52
Description: ETDRS-DRSS classifies diabetic retinopathy (DR) into 12 severity steps ranging from absence of retinopathy to advanced proliferative diabetic retinopathy (PDR). DRSS grades= 10 (DR absent) - 85 (very advanced PDR), DRSS 90 = ungradable. All DRSS values are converted into a 12-level scale, from 1 (DR absent) to 12 (very advanced PDR), allowing derivation of ≥2-step change from baseline for post-baseline assessment. A lower score represents less advanced diabetic retinopathy. The Cochran-Mantel Haenszel (CMH) method was used for analysis and weighted percentage of participants are estimated and reported in this outcome measure. Participants receiving supplemental treatments, prohibited therapy, or panretinal photocoagulation (PRP) were considered non-responders. Missing values not preceded by these intercurrent events were imputed using the last observation carried forward method. SD OCT= spectral-domain optical coherence tomography.
Time Frame: Baseline, Week 52
Population: ITT Population included all participants who were randomized. Participants were grouped according to treatment assigned at randomization.
Measure: Number; unit: percentage of participants
Arm/Group | PDS With Ranibizumab 100 mg/mL | Comparator Arm
Number analyzed (Participants) | 106 | 68
percentage of participants | 80.1 | 9.0
Statistical Analysis 1: Comparison: PDS With Ranibizumab 100 mg/mL vs Comparator Arm; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratification was done by baseline ETDRS-DRSS level (47 vs.53) & baseline intraretinal/subretinal fluid status on SD-OCT (present vs. absent); CMH Weighted Percentage Difference = 71.1, 95.04% CI 2-sided [61.0 to 81.2]

2. Secondary Outcome: Rate of Participants Developing a Vision-Threatening Complication or Center-involved Diabetic Macular Edema (CI-DME) Through Week 52
Description: A vision threatening complication is defined as proliferative DR (PDR) or anterior segment neovascularization (ASNV) or center-involved diabetic macular edema (CI-DME). CI-DME is defined as central foveal thickness (CST) ≥325 micrometres (μm) on spectral-domain optical coherence tomography (SD-OCT). Composite strategy (i.e., considered to be an event) was applied to participants who received supplemental or prohibited therapy or PRP in the study eye. The rate of participants was calculated using the Kaplan-Meier (KM) method.
Time Frame: From Baseline through Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | PDS With Ranibizumab 100 mg/mL | Comparator Arm
Number analyzed (Participants) | 106 | 68
percentage of participants | 7.1 | 47.0
Statistical Analysis 1: Comparison: PDS With Ranibizumab 100 mg/mL vs Comparator Arm; Test type: Superiority; p < 0.0001, Stratified Log-Rank; Stratified Hazard Ratio = 0.1, 95.04% CI 2-sided [0.1 to 0.3]; A stratified log-rank test was used for hypothesis testing comparing the PDS arm with the comparator arm. A Cox proportional hazards regression model (stratified) was used as a supportive analysis to estimate the Hazard ratio (HR)

3. Secondary Outcome: Rate of Participants Developing PDR or ASNV Through Week 52
Description: The KM method was used for analysis, and estimates are in terms of event rate. Composite strategy (i.e., considered to be an event) was applied to participants who received supplemental or prohibited therapy or PRP in the study eye.
Time Frame: From Baseline through Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | PDS With Ranibizumab 100 mg/mL | Comparator Arm
Number analyzed (Participants) | 106 | 68
percentage of participants | 1.0 | 42.4
Statistical Analysis 1: Comparison: PDS With Ranibizumab 100 mg/mL vs Comparator Arm; Test type: Superiority; p < 0.0001, Stratified Log-Rank; Stratified Hazard Ratio = 0.1, 95.04% CI 2-sided [0.1 to 0.1]; A stratified log-rank test was used for hypothesis testing comparing the PDS arm with the comparator arm. A Cox proportional hazards regression model (stratified) was used as a supportive analysis to estimate the HR

4. Secondary Outcome: Rate of Participants Developing CI-DME Through Week 52
Description: CI-DME is defined as CST ≥325 μm on SD-OCT. The KM method was used for analysis, and estimated in terms of event rate. Composite strategy (i.e., considered to be an event) was applied to participants who received supplemental or prohibited therapy or PRP in the study eye.
Time Frame: From Baseline through Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | PDS With Ranibizumab 100 mg/mL | Comparator Arm
Number analyzed (Participants) | 106 | 68
percentage of participants | 7.1 | 47.0
Statistical Analysis 1: Comparison: PDS With Ranibizumab 100 mg/mL vs Comparator Arm; Test type: Superiority; p < 0.0001, Stratified Log-Rank; Stratified Hazard Ratio = 0.1, 95.04% CI 2-sided [0.1 to 0.3]; [other analysis details as in outcome 3, analysis 1]

5. Secondary Outcome: Rate of Participants Developing a ≥ 2-Step Worsening From Baseline on the ETDRS-DRSS Through Week 52
Description: ETDRS-DRSS classifies diabetic retinopathy (DR) into 12 severity steps ranging from absence of retinopathy to advanced proliferative diabetic retinopathy (PDR). DRSS grades= 10 (DR absent) - 85 (very advanced PDR ), DRSS 90 = ungradable. All DRSS values are converted into a 12-level scale, from 1 (DR absent) to 12 (very advanced PDR), allowing derivation of ≥2-step change from baseline for post-baseline assessment. A lower score represents less advanced diabetic retinopathy. Composite strategy (i.e., considered to be an event) was applied to participants who received supplemental or prohibited therapy or PRP in the study eye. The rate of participants developing ≥ 2-step worsening on the ETDRS-DRSS was calculated using the KM method.
Time Frame: From Baseline through Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | PDS With Ranibizumab 100 mg/mL | Comparator Arm
Number analyzed (Participants) | 106 | 68
percentage of participants | 3.0 | 46.4
Statistical Analysis 1: Comparison: PDS With Ranibizumab 100 mg/mL vs Comparator Arm; Test type: Superiority; p < 0.0001, Stratified Log-Rank; Stratified Hazard Ratio = 0.1, 95.04% CI 2-sided [0.1 to 0.2]; [other analysis details as in outcome 3, analysis 1]

6. Secondary Outcome: Percentage of Participants With a ≥ 3-Step Improvement From Baseline on the ETDRS-DRSS at Week 52
Description: ETDRS-DRSS classifies diabetic retinopathy (DR) into 12 severity steps ranging from absence of retinopathy to advanced proliferative diabetic retinopathy (PDR). DRSS grades= 10 (DR absent) - 85 (very advanced PDR ), DRSS 90 = ungradable. All DRSS values are converted into a 12-level scale, from 1 (DR absent) to 12 (very advanced PDR), allowing derivation of ≥2-step change from baseline for post-baseline assessment. A lower score represents less advanced diabetic retinopathy. Participants receiving supplemental treatments, prohibited therapy, or panretinal photocoagulation (PRP) were considered non-responders. Missing values not preceded by these intercurrent events were imputed using the last observation carried forward method. Percentages are rounded off to the nearest decimal point.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | PDS With Ranibizumab 100 mg/mL | Comparator Arm
Number analyzed (Participants) | 106 | 68
percentage of participants | 15.1 | 0
Statistical Analysis 1: Comparison: PDS With Ranibizumab 100 mg/mL vs Comparator Arm; Test type: Superiority; p = 0.0003, Fisher Exact; Percentage Difference = 15.1, 95.04% CI 2-sided [8.3 to 21.9]

7. Secondary Outcome: Rate of Participants Developing a ≥ 3-Step Worsening From Baseline on the ETDRS-DRSS Through Week 52
Description: ETDRS-DRSS classifies diabetic retinopathy (DR) into 12 severity steps ranging from absence of retinopathy to advanced proliferative diabetic retinopathy (PDR). DRSS grades= 10 (DR absent) - 85 (very advanced PDR ), DRSS 90 = ungradable. All DRSS values are converted into a 12-level scale, from 1 (DR absent) to 12 (very advanced PDR), allowing derivation of ≥2-step change from baseline for post-baseline assessment. A lower score represents less advanced diabetic retinopathy. Composite strategy (i.e., considered to be an event) was applied to participants who received supplemental or prohibited therapy or PRP in the study eye. The rate of participants developing ≥ 3-step worsening on the ETDRS-DRSS was calculated using the KM method.
Time Frame: From Baseline through Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | PDS With Ranibizumab 100 mg/mL | Comparator Arm
Number analyzed (Participants) | 106 | 68
percentage of participants | 3.0 | 45.1
Statistical Analysis 1: Comparison: PDS With Ranibizumab 100 mg/mL vs Comparator Arm; Test type: Superiority; p < 0.0001, Stratified Log-Rank; Stratified Hazard Ratio = 0.1, 95.04% CI 2-sided [0.1 to 0.2]; [other analysis details as in outcome 3, analysis 1]

8. Secondary Outcome: Percentage of Participants With a ≥ 2-Step Improvement From Baseline on the ETDRS-DRSS Over Time
Description: ETDRS-DRSS classifies diabetic retinopathy (DR) into 12 severity steps ranging from absence of retinopathy to advanced proliferative diabetic retinopathy (PDR). DRSS grades= 10 (DR absent) - 85 (very advanced PDR), DRSS 90 = ungradable. All DRSS values are converted into a 12-level scale , from 1 (DR absent) to 12 (very advanced PDR), allowing derivation of ≥2-step change from baseline for post-baseline assessment. A lower score represents less advanced diabetic retinopathy.
Time Frame: Baseline up to Week 112
Reporting Status: Not Posted

9. Secondary Outcome: Percentage of Participants With a ≥ 3-step Improvement From Baseline on the ETDRS-DRSS Over Time
Description: ETDRS-DRSS classifies diabetic retinopathy (DR) into 12 severity steps ranging from absence of retinopathy to advanced proliferative diabetic retinopathy (PDR). DRSS grades= 10 (DR absent) - 85 (very advanced PDR ), DRSS 90 = ungradable. All DRSS values are converted into a 12-level scale , from 1 (DR absent) to 12 (very advanced PDR), allowing derivation of ≥2-step change from baseline for post-baseline assessment. A lower score represents less advanced diabetic retinopathy.
Time Frame: Baseline up to Week 112
Reporting Status: Not Posted

10. Secondary Outcome: Time to First Development of Either PDR, ASNV, or CI-DME
Time Frame: Baseline up to Week 112
Reporting Status: Not Posted

11. Secondary Outcome: Time to First Development of PDR or ASNV
Time Frame: Baseline up to Week 112
Reporting Status: Not Posted

12. Secondary Outcome: Time to First Development of CI-DME
Description: CI-DME is defined as CST ≥325 μm on SD-OCT.
Time Frame: Baseline up to Week 112
Reporting Status: Not Posted

13. Secondary Outcome: Time to First Development of a ≥ 2-Step Worsening From Baseline on the ETDRS-DRSS
Description: ETDRS-DRSS classifies diabetic retinopathy (DR) into 12 severity steps ranging from absence of retinopathy to advanced proliferative diabetic retinopathy (PDR). DRSS grades= 10 (DR absent) - 85 (very advanced PDR), DRSS 90 = ungradable. All DRSS values are converted into a 12-level scale, from 1 (DR absent) to 12 (very advanced PDR), allowing derivation of ≥2-step change from baseline for post-baseline assessment. A lower score represents less advanced diabetic retinopathy.
Time Frame: Baseline up to Week 112
Reporting Status: Not Posted

14. Secondary Outcome: Time to First Development of a ≥ 3-Step Worsening From Baseline on the ETDRS-DRSS
Description: as for outcome 13
Time Frame: Baseline up to Week 112
Reporting Status: Not Posted

15. Secondary Outcome: Change From Baseline in Best-Corrected Visual Acuity (BCVA) as Measured on the ETDRS Chart Over Time
Description: BCVA was measured at a starting test distance of 4 meters using a set of three Precision Vision^TM or Lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R). The BCVA letter score ranges from 0 to 100 (best score attainable), and a higher score indicates better visual acuity.
Time Frame: Baseline up to Week 112
Reporting Status: Not Posted

16. Secondary Outcome: Percentage of Participants Who Lost <15, <10 and <5 Letters in BCVA From Baseline Over Time
Description: BCVA was measured at a starting test distance of 4 meters using a set of three Precision VisionTM or Lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R). The BCVA letter score ranges from 0 to 100 (best score attainable), and a higher score indicates better visual acuity.
Time Frame: Baseline up to Week 112
Reporting Status: Not Posted

17. Secondary Outcome: Percentage of Participants With a BCVA Score of 69 Letters (20/40 Approximate Snellen Equivalent) or Better Over Time
Description: BCVA is measured using the ETDRS visual acuity chart starting at a test distance of 4 meters. The number of letters read correctly, Snellen fraction are converted to a decimal scale. There are 11 lines on a standard Snellen chart ranging from 0.1 (20/200) at worst to 2.0 (20/10) at best. 20/20 on the decimal scale is equal to 1.0. The higher the number of letters read correctly (higher number on the decimal scale), the better the vision (or visual acuity). The Snellen equivalent of 20/40 or better is 69 or more letters correctly read in the ETDRS chart.
Time Frame: Baseline up to Week 112
Reporting Status: Not Posted

18. Secondary Outcome: Change From Baseline in CST as Measured on SD-OCT Over Time
Description: CST is defined as the average thickness of the central 1 millimeter (mm) circle of the ETDRS grid centered on the fovea measured between the internal limiting membrane and the Bruch's membrane. CST is measured using spectral domain optical coherence tomography (SD-OCT). A central reading center graded the SD-OCT digital images. A negative change from baseline value represents a reduction in macular edema.
Time Frame: Baseline up to Week 112
Reporting Status: Not Posted

19. Secondary Outcome: Change From Baseline in Total Macular Volume (TMV) as Measured on SD-OCT Over Time
Description: Total macular volume in cubic millimeter (mm^3), is the calculated volume from the layers of the retina based off OCT imaging. TMV is measured using SD-OCT.
Time Frame: Baseline up to Week 112
Reporting Status: Not Posted

20. Secondary Outcome: Number of Participants With Ocular Adverse Events (AEs) and Severity of Ocular AEs in the PDS Arm
Description: An adverse event is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product,regardless of causal attribution.An adverse event can therefore be any unfavourable & unintended sign,symptom,or disease temporally associated with the use of a pharmaceutical product,whether considered related to the pharmaceutical product.Preexisting conditions which worsen during a study are also considered as adverse events.Ocular AEs are the events which are localized in the ocular region,graded according to the AE Severity Grading Scale as Mild:discomfort noticed,but no disruption of normal daily activity;Moderate:Discomfort sufficient to reduce or affect normal daily activity;Severe incapacitating with inability to work or to perform normal daily activity.Number of participants with ocular AEs in the study eye are reported in this outcome measure.As prespecified in the protocol, this outcome measure was applicable to participants in the PDS arm only.
Time Frame: From first dose of study drug through Week 52
Population: Safety Evaluable Population in the PDS arm included all participants randomized to PDS receiving at least one loading dose, or any participant who received the PDS implant prior to Week 52.
Measure: Count of Participants; unit: Participants
Arm/Group | PDS With Ranibizumab 100 mg/mL
Number analyzed (Participants) | 105
Participants
  Ocular AEs | 84
  Ocular AEs: Mild | 55
  Ocular AEs: Moderate | 21
  Ocular AEs: Severe | 8

21. Secondary Outcome: Number of Participants With Non-ocular AEs in the PDS Arm
Description: An adverse event is any untoward medical occurrence in a clinical investigation participant subject administered a pharmaceutical product, regardless of causal attribution. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events. As prespecified in the protocol, this outcome measure was applicable to participants in the PDS arm only.
Time Frame: From first dose of study drug through Week 52
Population: Safety Evaluable (SE) Population in the PDS arm included all participants randomized to PDS receiving at least one loading dose, or any participant who received the PDS implant prior to Week 52.
Measure: Count of Participants; unit: Participants
Arm/Group | PDS With Ranibizumab 100 mg/mL
Number analyzed (Participants) | 105
Participants | 59

22. Secondary Outcome: Number of Participants With At Least One Ocular Adverse Events of Special Interest (AESI) in the PDS Arm
Description: An AE is any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events. Ocular AESI include vitreous hemorrhage; endophthalmitis; retinal detachment; conjunctival retraction; conjunctival erosion; conjunctival bleb or conjunctival filtering bleb leak; hyphema; cataract; device dislocation. As prespecified in the protocol, this outcome measure was applicable to participants in the PDS arm only.
Time Frame: From first dose of study drug through Week 52
Population: SE Population in the PDS arm included all participants randomized to PDS receiving at least one loading dose, or any participant who received the PDS implant prior to Week 52.
Measure: Count of Participants; unit: Participants
Arm/Group | PDS With Ranibizumab 100 mg/mL
Number analyzed (Participants) | 105
Participants | 17

23. Secondary Outcome: Number of Participants With At Least One Ocular AESI During the Postoperative Period in the PDS Arm
Description: An AE is any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events. Ocular AESI include vitreous hemorrhage; endophthalmitis; retinal detachment; conjunctival retraction; conjunctival erosion; conjunctival bleb or conjunctival filtering bleb leak; hyphema; cataract; device dislocation. The ocular AESIs in the study eye were categorized based on onset as, Postoperative Period: onset within 37 days post initial implantation. As prespecified in the protocol, this outcome measure was applicable to participants in the PDS arm only.
Time Frame: From Day 1 to Day 37 Postoperative Period
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | PDS With Ranibizumab 100 mg/mL
Number analyzed (Participants) | 105
Participants
  Postoperative Period | 10
  Follow-up Period | 9

24. Secondary Outcome: Serum Concentration of Ranibizumab Observed Over Time
Time Frame: Baseline up to week 112
Reporting Status: Not Posted

25. Secondary Outcome: Pharmacokinetic (PK) Parameter Value Area Under the Concentration
Time Frame: At Baseline and multiple time points up to week 112
Reporting Status: Not Posted

26. Secondary Outcome: Minimum Serum Concentration (Cmin) of Ranibizumab Observed Over Time
Time Frame: Baseline up to week 112
Reporting Status: Not Posted

27. Secondary Outcome: Half-Life (t ½) of Ranibizumab Observed Over Time
Time Frame: Baseline up to Week 112
Reporting Status: Not Posted

28. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADAs) to Ranibizumab
Description: The numbers of ADA-positive participants at baseline and after drug administration were to be summarized for participants exposed to Ranibizumab. PDS patients who were ADA positive at the reference visit and ADA titer increased after implant; in this case, the titer of one or more samples collected after implant must be at least 4-fold greater than the titer of the reference visit sample. These patients are considered to have treatment-enhanced ADA responses.
Time Frame: Baseline up to Week 112
Reporting Status: Not Posted

29. Secondary Outcome: Number of Participants With Neutralizing Antibodies to Ranibizumab
Description: The numbers of neutralizing antibodies positive participants at baseline and after drug administration were to be summarized for participants exposed to Ranibizumab.
Time Frame: Baseline up to Week 112
Reporting Status: Not Posted

30. Secondary Outcome: Percentage of Participants Who do Not Undergo Supplemental Treatment With Intravitreal Ranibizumab Within Each Refill-Exchange Interval
Time Frame: Baseline up to Week 112
Reporting Status: Not Posted

31. Secondary Outcome: Percentage of Participants With At Least One AE Related to Study Device or Procedure in the PDS Arm
Description: An AE related to study device or procedure is defined as any adverse event related to the use of an investigational medical device. This includes any adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, operation, or any malfunction of the investigational medical device and any adverse event resulting from use error or from intentional misuse of the investigational medical device. PDS Device refers to the implant, insertion tool, initial fill needle, refill needle, and explant tool. PDS Procedure refers to the initial fill, implant insertion, refill-exchange, and explantation. As prespecified in the protocol, this outcome measure was applicable to participants in the PDS arm only. Percentages are rounded off to the nearest decimal point.
Time Frame: From first dose of study drug through Week 52
Population: as for outcome 22
Measure: Number; unit: percentage of participants
Arm/Group | PDS With Ranibizumab 100 mg/mL
Number analyzed (Participants) | 105
percentage of participants | 70.5

32. Secondary Outcome: Percentage of Participants With Serious Adverse Effects Related to Study Device or Procedure in the PDS Arm
Description: An AE related to study device or procedure is defined as any AE related to the use of an investigational medical device & includes any AE resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, operation, or any malfunction of the investigational medical device & any AE resulting from use error or from intentional misuse of the investigational medical device. PDS refers to the implant, insertion tool, initial fill needle, refill needle & explant tool. PDS procedure refers to the initial fill, implant insertion, refill-exchange, & explantation. Any AE related to study device or procedure that resulted in any of a serious AE such as death, life-threatening illness or injury or permanent impairment of a body structure or a body function was considered serious. As prespecified in the protocol, this outcome measure was applicable to participants in the PDS arm only. Percentages are rounded off to the nearest decimal point.
Time Frame: From Day 1 up to Week 52
Population: as for outcome 22
Measure: Number; unit: percentage of participants
Arm/Group | PDS With Ranibizumab 100 mg/mL
Number analyzed (Participants) | 105
percentage of participants | 1.0

33. Secondary Outcome: Percentage of Participants With Absence of Intraretinal Fluid, Subretinal Fluid or Both Over Time
Description: Absence of intraretinal fluid and subretinal fluid are measured in the central 1 mm subfield on SD-OCT. Percentages are rounded off to the nearest decimal point.
Time Frame: Baseline up to Week 112
Reporting Status: Not Posted

34. Secondary Outcome: Percentage of Participants Who Report Preferring PDS Treatment to Intravitreal Ranibizumab Treatment, as Measured by the PDS Patient Preference Questionnaire (PPPQ) at Week 52
Description: The PPPQ is a 3-item questionnaire that captures a participant's preference for treatment (PDS or intravitreal injections), the strength of their preference (very strong, fairly strong, and not very strong) and the reasons for their preference (less worry or nervousness, requires less time for treatment, less discomfort, fewer treatments and other reason). As prespecified in the protocol, this outcome measure was applicable to participants in the PDS arm only. Percentages are rounded off to the nearest decimal point.
Time Frame: Week 52
Population: ITT Population included all participants who were randomized. Overall number analyzed is the number of participants who completed the questionnaire.
Measure: Number; unit: percentage of participants
Arm/Group | PDS With Ranibizumab 100 mg/mL
Number analyzed (Participants) | 94
percentage of participants | 76.6

35. Secondary Outcome: Number of Participants With Device Deficiencies
Description: A device deficiency is defined as any inadequacy with respect to labeling, identity, quality, durability, reliability, usability, safety, or performance of an investigational device, including malfunctions, use errors, or inadequacy in information supplied by the manufacturer. As prespecified in the protocol, this outcome measure was applicable to participants in the PDS arm only and device deficiencies were to be recorded in the electronic capture system (EDC) after implementation of protocol Version 2 (i.e., for participants implanted after 14 June 2021).
Time Frame: Baseline up to Week 52
Population: SE Population in the PDS arm included all participants randomized to PDS receiving at least one loading dose, or any participant who received the PDS implant prior to Week 52. Overall number analyzed is the number of participants implanted after 14 June 2021.
Measure: Count of Participants; unit: Participants
Arm/Group | PDS With Ranibizumab 100 mg/mL
Number analyzed (Participants) | 47
Participants | 9

ADVERSE EVENTS:
Time Frame: From study start through primary completion date (up to Week 52)
Description: All-cause mortality:ITT.Serious & other AEs:SE Population.Per-protocol,AE collection began after 1st study treatment(ST) besides limited key exceptions;ST was mandatory for PDS arm.In Comparator arm (CA),27of 68 participants received ST & reported all AEs; safety follow-up for them varied through Week 52(8-356 days). The remaining 41 participants in CA were not required to report all AEs, precluding a complete AE analysis.AEs for all implanted participants will be provided at the final analysis.
Arm/Group | PDS With Ranibizumab 100 mg/mL
All-Cause Mortality (participants affected / at risk) | 0/106
Serious Adverse Events (participants affected / at risk) | 17/105
Other Adverse Events (participants affected / at risk) | 89/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PDS With Ranibizumab 100 mg/mL (N=105)
Acute myocardial infarction (Cardiac disorders) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 3 (3)
Coronary artery disease (Cardiac disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1) — For this AE, the number of participants and events reported per term are combined totals of AEs that occurred in the study eye or the fellow eye.
Diabetic retinopathy (Eye disorders) | 1 (1) — For this AE, the number of participants and events reported per term are combined totals of AEs that occurred in the study eye or the fellow eye.
Ocular hypertension (Eye disorders) | 1 (1) — For this AE, the number of participants and events reported per term are combined totals of AEs that occurred in the study eye or the fellow eye.
Retinal artery occlusion (Eye disorders) | 1 (1) — For this AE, the number of participants and events reported per term are combined totals of AEs that occurred in the study eye or the fellow eye.
Retinal detachment (Eye disorders) | 1 (1) — For this AE, the number of participants and events reported per term are combined totals of AEs that occurred in the study eye or the fellow eye.
Vitreous haemorrhage (Eye disorders) | 1 (1) — For this AE, the number of participants and events reported per term are combined totals of AEs that occurred in the study eye or the fellow eye.
Constipation (Gastrointestinal disorders) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PDS With Ranibizumab 100 mg/mL (N=105)
Cataract (Eye disorders) | 6 (8) — For this AE, the number of participants and events reported per term are combined totals of AEs that occurred in the study eye or the fellow eye.
Conjunctival haemorrhage (Eye disorders) | 79 (93) — For this AE, the number of participants and events reported per term are combined totals of AEs that occurred in the study eye or the fellow eye.
Conjunctival hyperaemia (Eye disorders) | 12 (12) — For this AE, the number of participants and events reported per term are combined totals of AEs that occurred in the study eye or the fellow eye.
Conjunctival oedema (Eye disorders) | 10 (10) — For this AE, the number of participants and events reported per term are combined totals of AEs that occurred in the study eye or the fellow eye.
Diabetic retinal oedema (Eye disorders) | 6 (7) — For this AE, the number of participants and events reported per term are combined totals of AEs that occurred in the study eye or the fellow eye.
Diabetic retinopathy (Eye disorders) | 7 (8) — For this AE, the number of participants and events reported per term are combined totals of AEs that occurred in the study eye or the fellow eye.
Eye pain (Eye disorders) | 9 (15) — For this AE, the number of participants and events reported per term are combined totals of AEs that occurred in the study eye or the fellow eye.
Foreign body sensation in eyes (Eye disorders) | 9 (9) — For this AE, the number of participants and events reported per term are combined totals of AEs that occurred in the study eye or the fellow eye.
Iritis (Eye disorders) | 10 (10) — For this AE, the number of participants and events reported per term are combined totals of AEs that occurred in the study eye or the fellow eye.
Ocular hypertension (Eye disorders) | 7 (9) — For this AE, the number of participants and events reported per term are combined totals of AEs that occurred in the study eye or the fellow eye.
Punctate keratitis (Eye disorders) | 10 (14) — For this AE, the number of participants and events reported per term are combined totals of AEs that occurred in the study eye or the fellow eye.
Vitreous detachment (Eye disorders) | 9 (10) — For this AE, the number of participants and events reported per term are combined totals of AEs that occurred in the study eye or the fellow eye.
Vitreous haemorrhage (Eye disorders) | 14 (14) — For this AE, the number of participants and events reported per term are combined totals of AEs that occurred in the study eye or the fellow eye.
COVID-19 (Infections and infestations) | 16 (16)
Sinusitis (Infections and infestations) | 7 (7)
Headache (Nervous system disorders) | 9 (11)
Hypertension (Vascular disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-06-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT04503551/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-03): https://cdn.clinicaltrials.gov/large-docs/51/NCT04503551/SAP_001.pdf